CLINICAL TRIAL: NCT01941602
Title: A Comparative Study of Prophylactic Enoxaparin Routinely Administered Preoperative for Prevention of Venous Thromboembolism in Meningioma Surgery - an Acceptable Risk-benefit Ratio?
Brief Title: A Comparative Study of Prophylactic Anticoagulation in Meningioma Surgery
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); University Hospital of North Norway (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/884
Record Dates: First submitted 2013-09-02; First posted 2013-09-13 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Meningioma
Keywords: surgery; enoxaparin; venous thromboembolism; perioperative care
MeSH Terms: conditions — Meningioma; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prophylactic: Prophylactic treatment with drugs to prevent venous thromboembolism in patients operated with open surgery for intracranial meningioma at the Department of neurosurgery at Karolinska Hospital, Stockholm, Sweden
  Interventions: Drug: prophylactic enoxaparin
- non-prophylactic: No use of prophylactic treatment with drugs to prevent venous thromboembolism in patients operated with open surgery for intracranial meningioma at the Departments of neurosurgery at University Hospital North Norway (UNN) and St.Olavs University Hospital (Tromsø and Trondheim respectively, both Norway)
  Interventions: Procedure: non-prophylactic

INTERVENTIONS:
Drug: prophylactic enoxaparin — enoxaparin had been prescribed at a dose of 40 mg (once daily) from the evening before surgery until patients were well mobilized. Also, at the time of surgery compression stockings were used, as well as a sequential compression device (SCD) until the morning after or longer if mobilization was delayed
  Groups: prophylactic
Procedure: non-prophylactic — no pharmacological prophylaxis for venous thromboembolism (VTE) had been used routinely. Occasionally, with delayed mobilization, a low-dose low molecular weight heparin (LMWH) had been prescribed. SCD had been used at increased frequency, and is today considered routine.
  Groups: non-prophylactic

SUMMARY:
The aim of the study is to compare different strategies for prevention of venous thromboembolism related to intracranial meningioma surgery. The investigators identified three hospitals where two have a very restrictive approach with respect to anticoagulant therapy while at the third hospital the use of anticoagulation the day before surgery was initiated as routine prophylaxis.

Based on this "natural experiment" it will be explored whether the use of anticoagulant prophylaxis is associated with reduced risk of venous thromboembolism and/or associated with increased risk of postoperative hemorrhage as compared to the 2 cohorts where this intervention were absent.

ELIGIBILITY:
Inclusion Criteria:

* First included patient 1.january 2007 and latest included patient 1.july 2013 (allows for 30 day follow up with respect to morbidity)
* Histological verification of a meningioma (of any grade) from the current surgery

Exclusion Criteria:

* Intracranial surgery or venous thromboembolism the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having had surgical treatment for intracranial meningioma in Norway (St Olavs University Hospital, Trondheim, and University Hospital North Norway, Tromsø) and Sweden (Karolinska University Hospital, Stockholm).
Sampling Method: Non-Probability Sample
Enrollment: 979 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
frequencies of venous thromboembolism | 30 days

SECONDARY OUTCOMES:
frequencies of hematomas in need of reoperation or that significantly alters subsequent care | 30 days
  frequencies of hematomas in need of reoperation or that significantly alters subsequent care (e.g. intensive care unit or other intensified treatment based on postoperative intracranial hemorrhage)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jacob Stovner, MD PhD, Study Director — St. Olavs Hospital
Locations (3):
- Norway (2):
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Sjavik K, Bartek J Jr, Solheim O, Ingebrigtsen T, Gulati S, Sagberg LM, Forander P, Jakola AS. Venous Thromboembolism Prophylaxis in Meningioma Surgery: A Population-Based Comparative Effectiveness Study of Routine Mechanical Prophylaxis with or without Preoperative Low-Molecular-Weight Heparin. World Neurosurg. 2016 Apr;88:320-326. doi: 10.1016/j.wneu.2015.12.077. Epub 2015 Dec 31. PMID 26746334